CLINICAL TRIAL: NCT05696808
Title: Effects of Indian Foods and Ayurvedic Drugs on Healthy and Diseased Liver
Brief Title: Effect of Indian Hepatoprotective Diet in Reversibility of NAFLD
Acronym: NAFLDNutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-NAFLD
Record Dates: First submitted 2023-01-14; First posted 2023-01-25 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome | interventions — Diet, Western

STUDY DESIGN:
Intervention Model Description: All the variables would be studied before and after intervention with indian hepatoprotective diet (IHPD) in 60 patients with NAFLD and 60 healthy individuals on Western diet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indian hepatoprotective diet (IHPD) (Experimental): The intervention is planned as a supervised dietary supplementation, with a goal of restricting the calorie intake to 25 Kcal/Kg BW/day, with a protein intake of 1 gm/Kg BW/day i.e., around 15 % of total calories from protein, 35% from fats and 50% from carbohydrates. Major portion of the carbohydrates is vegetables, fruits and then cereals (high fiber cereals), more amount of tomato and amla at least 200 gm in a day, protein requirements are met by mainly legumes like chick pea black - (kala chana) and moong sprouts besides dals. Lean meats and egg whites would be allowed as the non-vegetarian source. Milk products used are only milk and buttermilk, curd (excluding paneer). Major source of oil would be mustard oil only.
  Interventions: Dietary Supplement: IHPD
- Western Diet (Active Comparator): The intervention is planned with a goal of restricting the calorie intake to 40 Kcal/Kg BW/day, around 10-15 % of total calories from protein, 30-35% from fats and 55-60% from carbohydrates. Major portion of the carbohydrates is Western fast food comprising of pizza and burger, French fries, sweets, muffins, cakes, chocolates, sugar sweetened beverages.
  Interventions: Dietary Supplement: Western Diet

INTERVENTIONS:
Dietary Supplement: IHPD — The intervention is planned as a supervised dietary supplementation, with a goal of restricting the calorie intake to 25 Kcal/Kg BW/day, with a protein intake of 1 gm/Kg BW/day i.e., around 15 % of total calories from protein, 35% from fats and 50% from carbohydrates. Major portion of the carbohydrates is vegetables, fruits and then cereals (high fiber cereals), more amount of tomato and amla at least 200 gm in a day, protein requirements are met by mainly legumes like chick pea black - (kala chana) and moong sprouts besides dals. Lean meats and egg whites would be allowed as the non-vegetarian source. Milk products used are only milk and buttermilk, curd (excluding paneer). Major source of oil would be mustard oil only.
  Arms: Indian hepatoprotective diet (IHPD)
Dietary Supplement: Western Diet — The intervention is planned with a goal of restricting the calorie intake to 40 Kcal/Kg BW/day, around 10-15 % of total calories from protein, 30-35% from fats and 55-60% from carbohydrates. Major portion of the carbohydrates is Western fast food comprising of pizza and burger, French fries, sweets, muffins, cakes, chocolates, sugar sweetened beverages.
  Arms: Western Diet

SUMMARY:
The modality of lifestyle modification including low calorie diets along with normal protein and moderate physical activity is the safest standard medical treatment for NAFLD in general. There are many benefits of weight loss to the patients with NAFLD. Besides the improvement in the features of metabolic syndrome, weight loss with IHPD would certainly improve the overall vitality and well being of the patients. The results of study will help to delineate a protocolized care for the management of NAFLD with metabolic syndrome thus helping other patients also in the future.

DETAILED DESCRIPTION:
There is a strong link between food items, gut microbiota (GM), liver fat and development of various non-communicable diseases (NCDs). The incidence of NCDs is rapidly increasing globally. The GM is considered an organ by itself and any alterations in its composition or functioning are likely to be associated with different NCDs, including cancers. The core to most of the NCDs is increased fat in the liver and the non-alcoholic fatty liver disease (NAFLD). The highly variable natural history of NAFLD reflects the current incomplete understanding of the pathobiology of the disease. The strongest risk factors for NAFLD/NASH are unhealthy food items and their metabolites which affect the host and the gut microbiota.

Traditional Indian food items are known to have strong influence on liver and production of healthy bile, the 'Pitta'. The influence and health worthiness of various indigenous food items has not been scientifically evaluated. Their role in health and disease would not only help in prevention but also management of multiple non-communicable diseases. This information could also make a change in the social and behavioural attitudes of Indians

The proposed project would, therefore, undertake work on the following broad areas:

1. Effects of conventional Indian foods as hepatoprotective agents, producers of 'healthy' bile and stimulating liver regeneration.
2. Food constituents as therapeutic agents by changing dysbiotic gut microbiota to healthy microbiota, reduction in hepatic fat and inflammation, improving metabolic health (reducing sugar, cholesterol, etc.) and reduction in liver fibrosis

ELIGIBILITY:
Inclusion Criteria:

1. Patients recently diagnosed (<3 months)diagnosed on the basis of ultrasound and /or liver transient eleastography (controlled attenuation parameter; CAP >250)
2. Having components of metabolic syndrome like Hyperglycemia, central obesity, hypertension, hypertriglyceridemia, and low HDL cholesterol levels).

Exclusion Criteria:

1. Pregnant & lactating women
2. Age <18 and >55 years
3. Individuals who had been hospitalised with complications of Diabetes mellitus, Chronic Kidney disease, Hypertension in the previous 6 months
4. Those with intake of antibiotics within last month
5. Seriously ill and bed ridden patients
6. Patients with viral hepatitis
7. Patients with significant alcohol consumption (regular consumption of > 10g per day for females and > 20g/d in males),
8. Patients having chronic inflammatory bowel disease or any chronic and autoimmune diseases will be excluded
9. Patients with NAFLD with associated hypertriglyceridemia requiring administration of statins.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-01-13 (Estimated)

PRIMARY OUTCOMES:
To study the effectiveness of Indian Hepatoprotective Diet (IHPD) in hepatic steatosis in patients with NAFLD index in patients with NAFLD | 1 month
  Hepatic steatosis index will be assessed by controlled attenuation parameter (CAP) score.

SECONDARY OUTCOMES:
To study the effectiveness of IHPD on Hyperglycemia (Fasting blood sugar) in patients with NAFLD | 1 month
  Hyperglycemia will checked by fasting blood sugar>110mg/dl
To study the effectiveness of IHPD on central obesity (waist circumference) in patients with NAFLD | 1 month
  Central obesity will be measured by waist circumference in cm
To study the effectiveness of IHPD on hypertension (BP) in patients with NAFLD | 1 month
  Hypertension will be checked by observing blood pressure>120/80
To study the effectiveness of IHPD on hypertriglyceridemia in patients with NAFLD | 1 month
  Hypertriglyceridemia will be checked by raised cholestrol and triglycerides.
To study the effectiveness of IHPD in reducing body weight in patients with NAFLD | 1 month
  Weight will be checked in kg with the help of weihing machine
To study the effectiveness of IHPD on gut microbiota in patients with NAFLD | 1 month
  Gut microbiota will be assessed by 16S

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Shiv Kr Sarin, MD, DM, FNA, Principal Investigator — Institute of Liver and Biliary Sciences, New Delhi, India
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No